CLINICAL TRIAL: NCT04195178
Title: Understanding the Cognition and Decision Making of Community Anesthesiologists in Their Management of End-of-case Neuromuscular Blockade: a Mixed Methods Study
Brief Title: Understanding the Cognition and Decision Making of Community Anesthesiologists
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: University of Pittsburgh (Other); The Cooper Health System (Other)
Responsible Party: Principal Investigator, Matthew Weinger, Professor, Vanderbilt University Medical Center
Other Study IDs: 181711
Record Dates: First submitted 2019-11-30; First posted 2019-12-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2024-02

CONDITIONS: Neuromuscular Blockade

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Anesthesia Providers: Clinically active anesthesia providers

SUMMARY:
The investigators are interested in studying why experienced clinicians make specific decisions regarding the monitoring of patients' physiological states and why clinicians might make decisions that are contrary to current best practices or known evidence. More generally, the program objective is to refine and validate a novel methodology to delineate clinicians' decision-making strategies. More specifically, the investigators will study the decision to reverse neuromuscular blockade at the end of an anesthetic. This clinical decision will be studied in this project because: 1) it has been well documented that a substantial percentage of practitioners do not follow best practices; 2) the variables are relatively circumscribed and well described; and 3) it can be framed as a binary decision.

The investigators propose to conduct an observational mixed-methods study developing and using clinical vignettes and cognitive interviews to better understand the decision-making approaches and preferences of clinically active anesthesia providers with regard to their decision-making during clinical anesthesia cases. After developing clinical vignettes and related questions, the investigators will first obtain detailed demographic and clinical practice variables from the participants via a survey. Participants will then review multiple vignettes that present different clinical situations that focus on decisions to reverse neuromuscular blockade and/or extubate the patient. Each participant will provide their decisions for each vignette. The investigators will then conduct an audiotaped interview, using cognitive task analysis methods, to ascertain the factors that played a role in these decisions.

DETAILED DESCRIPTION:
The investigators propose to conduct a 3-site prospective observational mixed-methods study using clinical vignettes and cognitive interviews to better understand the decision making approaches and preferences of practicing community anesthesiologists with regard to the management of non-depolarizing neuromuscular blockade (NMB) at the end of general endotracheal anesthesia cases.

The objectives of this initial study is to begin to understand:

1. When and why do community anesthesiologists choose to reverse NMB?
2. What are the decision preferences of community anesthesiologists with regard to their decisions to reverse NMB, and what are the clinician and clinical case factors that influence those decisions?
3. What are the operational knowledge gaps of anesthesia professionals with regard to their ability to follow best-practice evidence for the reversal of NMB? More generally, the program objective is to refine and validate a novel methodology to delineate clinicians' decision making strategies and triggers.

2.1.2. Study Hypotheses

For this initial study, the investigators hypothesize that:

1. There will be a significant distribution of clinical variables across community anesthesiologists' decision to reverse NMB.
2. There will be measurable differences in participant demographics and practice attributes between those who closely follow evidence-based expectations for reversal of NMB and those who do not. The investigators expect community practitioners who do not reverse NMB in accordance with current best evidence to be older, to not be fellowship trained or subspecialty certified, and to practice in lower acuity settings.

This will be a remotely conducted national prospective observational simulation study of 36 experienced community anesthesiologists using a clinical vignette and cognitive interviews to better understand the decision making approaches and preferences of practicing community anesthesiologists with regard to the management of neuromuscular blockade (NMB) at the end of general endotracheal anesthesia cases.

Cognitive interview transcript coders and analysts will be blinded to the identity and attributes of the participants.

ELIGIBILITY:
Inclusion Criteria:

* Clinically active experienced anesthesia providers

Exclusion Criteria:

* Anesthesia providers who are no longer practicing or clinically active

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinically active anesthesia providers
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2023-08-03 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Average Decision Thresholds: Pharmacological measure of neuromuscular blocking drug effect | 10 minutes
  The average decision threshold is the average across all participant's decision threshold for this measure. The decision threshold is calculated by sequentially varying values of the pharmacological variables (i.e., doses and timing) within the context of a clinical scenario. Each participant's decision threshold is the equivalent of an ED50 or a MAC value (i.e., the equipoise point for their clinical decision based on that variable).
Average Decision Thresholds: Muscle strength | 10 minutes
  The average decision threshold is the average across all participant's decision threshold for this measure. The decision threshold is calculated by sequentially varying values of muscle strength within the context of a clinical scenario. Each participant's decision threshold is the equivalent of an ED50 or a MAC value (i.e., the equipoise point for their clinical decision based on that variable).
Average Decision Thresholds: Respiratory parameters | 10 minutes
  The average decision threshold is the average across all participant's decision threshold for this measure. The decision threshold is calculated by sequentially varying values of the respiratory parameters (i.e., variables contributing to minute ventilation) within the context of a clinical scenario. Each participant's decision threshold is the equivalent of an ED50 or a MAC value (i.e., the equipoise point for their clinical decision based on that variable).

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided